CLINICAL TRIAL: NCT04664140
Title: Angio-based Quantitative Flow Ratio Virtual PCI Versus Conventional Angio-guided PCI in the Achievement of an Optimal Post-PCI QFR
Brief Title: QFR-based Virtual PCI Versus Angio-guided PCI
Acronym: AQVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Full Professor of Cardiology, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1021/2020/Sper/AOUFe
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Percutaneous Coronary Intervention; Coronary Physiology
Keywords: angio-based FFR; percutaneous coronary intervention

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: The core-laboratory will be blinded to patients randomization during the adjudication of the endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QFR-based virtual PCI (Experimental): Before starting PCI, the operator must acquire QFR angiographic projections after nitroglycerin administration at 15 frames/second. Angiographic projections should be at least 25 apart, aiming for minimal vessel foreshortening and minimal vessel overlap. In agreement with previous studies, operators follow a table of recommended projection angles. Afterwards, online QFR analysis must be performed. The tool "residual vessel QFR" should be used to anticipate the result of stenting (virtual PCI) by placing the proximal (p) and distal (d) marker in order to obtain a post-PCI QFR ≥0.90. then, the operator has to implant one or more stents following the pre-PCI plan and utilizing the QFR and angio to place the stent(s) according to the virtual PCI plan. Post-dilation with non-compliant (NC) balloon is strongly suggested. Blinded QFR projections must be obtained after PCI.
  Interventions: Other: QFR-based virtual PCI
- Angiography-based PCI (Active Comparator): Invasive coronary angiography and PCI are performed following best local practices. Post-dilation with a noncompliant balloon is strongly suggested. Blinded QFR projections must be obtained before and after PCI.
  Interventions: Other: angiography-based PCI

INTERVENTIONS:
Other: QFR-based virtual PCI — Procedural planning of PCI based on the pullback trace given by the QFR systems in order to obtain an optimized functional result after PCI
  Other Names: angio-FFR based virtual PCI
  Arms: QFR-based virtual PCI
Other: angiography-based PCI — PCi according to international guidelines, local protocols and practice
  Other Names: angio-based PCI
  Arms: Angiography-based PCI

SUMMARY:
A significant portion of patients continue to experience both adverse events and symptoms after angiographically successful PCI. Beyond different underlying mechanisms non-related to epicardial disease (vasospasm, microcirculatory dysfunction), several recent studies have shown that in at least 15-20% of PCIs, a prognostically meaningful ischemia, detected with different coronary physiology tools, is present at the end of a successful angiography-guided PCI. In addition, physiology is able to discriminate the underlying reason causing the suboptimal functional result, namely: i) in-stent drop; ii) focal drop outside stent; iii) diffuse disease.

However, the use of post-PCI physiology is still very low, even when it is utilized pre-PCI to set the indication for stenting. Lack of dedicated randomized clinical trials and procedural lengthening and increase in side effects are at the basis of this underutilization.

In addition, the ideal tool should allow to plan the intervention in advance rather than to assess the results afterwards. To this hand, QFR is particularly appealing, among available physiology tools, because it does not need wire or adenosine and allows: i) identification of disease mechanism; ii) co-registration with angiography; iii) pre-PCI planning with residual vessel QFR value according to a pre-specified treatment.

Taken all this characteristics together, QFR is the ideal technology for virtual PCI.

The hypothesis of the present investigation is that a procedural planning based on QFR (virtual PCI) is able to reduce the rate of patients with post-PCI suboptimal functional result, that has been found to correlate with prognosis in our earlier study, if compared to the traditional angio-guided PCI.

DETAILED DESCRIPTION:
Post-percutaneous coronary intervention (PCI) physiology The results of functional assessment performed after percutaneous coronary intervention (PCI) taught us that a "successful" angiography-guided PCI is often suboptimal in terms of physiology and that physiology result after PCI is closely linked to outcome. Yet, post-PCI physiology is rarely utilized in clinical practice, being employed in less than 10% of lesions investigated with physiology pre-PCI. Reasons for the low use of functional assessment post-PCI and for subsequent intervention are manifold. First, physiology is actually used after PCI only in cases where it was utilized pre-PCI. Second, randomized clinical trials (RCT) addressing the use of physiology to assess PCI results have not been performed, therefore clear instructions and cutoffs for its use are lacking. Third, when fractional flow reserve (FFR) is measured, the need to administer adenosine several times during the same procedure results in increased procedure time, cost and adverse side effects. Fourth, in case of a post-PCI suboptimal functional result, it may be difficult to ascertain the underlying cause.

New indices and tools have been developed in an effort to overcome barriers to the widespread adoption of functional assessment. Non-hyperaemic pressure indices (NHPI) including, resting distal to aortic coronary pressure ratio (Pd/Pa), and other resting indices have enabled functional evaluation without pharmacological arteriolar vasodilation, while angiography-based functional assessment have eliminated the need for a dedicated pressure wire.

Importantly, these newer tools may allow operators to understand the mechanism underlying an abnormal physiology value after angiographically successful intervention. In fact, the real novelty related to their development is the shift from a binary interpretation of physiology (positive/negative) to a quantitative site-specific one. For these reasons, they are extremely appealing post-PCI and several studies have been recently conducted to validate them in this setting.

Quantitative flow ratio (QFR) In particular, quantitative flow ratio (QFR) is an angiographically-derived estimate of FFR developed as an alternative to wire-based intracoronary physiology. One advantage of angio-based FFR systems is allowing the generation of a pullback curve and discrimination of the physiological contribution of each single lesion as well as diagnosis of diffuse disease. The value of QFR to assess the functional results of PCI has been tested in the prospective Angio-Based Fractional Flow Reserve to Predict Adverse Events After Stent Implantation (HAWKEYE) study. Seven hundred fifty-one vessels in 602 patients undergoing angiographically satisfactory second-generation drug eluting stent (DES) implantation were analyzed. At the end of the procedure, the operator acquired projections for QFR computation performed offline by an independent core laboratory. Receiver operating characteristic (ROC) curve analysis identified a post-PCI QFR best cut-off of <0.90 (area under the curve 0.77; 95% confidence interval [CI]: 0.74-0.80; p< 0.001). After correction for potential confounding factors, post-PCI QFR<0.90 was associated with a 3-fold increase in risk for the vessel-oriented composite endpoint at 2 years (HR: 2.91; 95% CI 1.63-5.19; p< 0.001). Further, a very important finding of the HAWKEYE study was the demonstration that QFR could discriminate among different coronary artery disease (CAD) patterns. In vessels with suboptimal functional result, the site of the QFR drop was in-stent in 13% of the cases, while a focal drop outside the stent was identifiable in 32% of the cases. Thirty-four percent of vessels showed diffuse disease, while in 21% a combination of the aforementioned possibilities was present. It is important to note that QFR analyzability depends on quality of angiography and it is feasible in around 80% of the cases. Moreover, QFR is not applicable in specific lesion subsets such as left main, bifurcation and ostial lesions.

Virtual PCI The inherent limit of post-PCI physiology is to add measurement and consequent actions after the end of a procedure that has been deemed successful by the same operator who is performing it. In addition, it is associated with the increase in procedural time and costs. Thus, a broad application of post-PCI physiology, although clinically meaningful, is implausible.

On the contrary, the systematic application of QFR before stenting to simulate PCI results according to different treatment strategies (virtual PCI) would be an interesting alternative to achieve a fully physiology guided procedure.

The advantages of a virtual PCI strategy based on QFR application are:

* QFR is a simple tool, based on what the operator already performs before PCI (namely two perpendicular angiographic projections) and not requiring wire or adenosine.
* It enables to obtain a full physiologic map of the vessel with a point-by-point detailed information of the functional impact of a given stenosis.
* It is possible to simulate the treatment of one or more lesions (virtual PCI) in order to estimate the final functional value post-PCI.

Then, virtual PCI based on QFR utilization would not increase procedural time or costs and could obtain an optimal post-PCI physiology result in most cases. The "Angio-based Quantitative flow ratio Virtual PCI versus Conventional Angio-guided PCI in the achievement of an optimal post-PCI QFR" (AQVA) trial is the first step toward this direction and will be the basis for a bigger study focused on hard clinical endpoints.

OBJECTIVES

To evaluate:

* The rate of lesions with a final post-PCI QFR≥0.90 in patients treated with the QFR virtual PCI versus patients treated with an angiography-based PCI.
* The rate of vessel-oriented composite endpoint (VOCE), defined as the composite of vessel-related cardiovascular death, vessel-related myocardial infarction (MI), and ischemia-driven target vessel revascularization (TVR).

SAMPLE SIZE CALCULATION

In the HAWKEYE trial population, 16% of lesions presented a post-PCI QFR <0.90 after an angio-guided PCI. In one third of these lesions, low post-PCI QFR was due to diffuse disease. Therefore, the investigators hypothesize that a procedural plan with QFR could be able to reduce the rate of lesions with QFR<0.90 by two thirds. Considering that some of the lesions with focal disease could also present diffuse disease, the investigators can realistically estimate a reduction by 60% with virtual-PCI. Therefore, 300 patients are required to have a 80% chance of detecting, as significant at the 5% level, an increase in the percentage of patient achieving a post-PCI QFR≥0.90 from 84% in the angio-guided group to 94% in the virtual PCI group.

ELIGIBILITY:
Inclusion Criteria:

* Indication to PCI for either acute or chronic coronary syndrome
* Signed informed consent

Exclusion Criteria:

* Planned surgical revascularization
* Prior Coronary Artery Bypass Graft (CABG) Surgery
* Culprit lesion of STEMI or NSTEMI
* Clinical or angiographic features limiting QFR computation:
* Left main or ostial right coronary artery
* Atrial fibrillation
* Ongoing ventricular arrhythmias
* Significant and persistent tachycardia
* Revascularization of a chronic total occlusion
* Non-cardiovascular co-morbidity reducing life expectancy to < 1 year
* Any factor precluding 1-year follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
post-PCI QFR | end of the procedure
  proportion of patients with a final post-PCI QFR result ≥0.90

SECONDARY OUTCOMES:
vessel-oriented composite endpoint (VOCE) | 1 year
  composite of vessel-related cardiovascular death, vessel-related MI, and ischemia-driven target vessel revascularization (TVR)

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - University Hospital of Ferrara, Cona, Ferrara
  - University Hospital Federico II, Napoli
  - Azienda Ospedaliera Santa Maria, Reggio Emilia

REFERENCES:
- [Background] Biscaglia S, Tebaldi M, Brugaletta S, Cerrato E, Erriquez A, Passarini G, Ielasi A, Spitaleri G, Di Girolamo D, Mezzapelle G, Geraci S, Manfrini M, Pavasini R, Barbato E, Campo G. Prognostic Value of QFR Measured Immediately After Successful Stent Implantation: The International Multicenter Prospective HAWKEYE Study. JACC Cardiovasc Interv. 2019 Oct 28;12(20):2079-2088. doi: 10.1016/j.jcin.2019.06.003. Epub 2019 Sep 25. PMID 31563688
- [Background] Jeremias A, Davies JE, Maehara A, Matsumura M, Schneider J, Tang K, Talwar S, Marques K, Shammas NW, Gruberg L, Seto A, Samady H, Sharp A, Ali ZA, Mintz G, Patel M, Stone GW. Blinded Physiological Assessment of Residual Ischemia After Successful Angiographic Percutaneous Coronary Intervention: The DEFINE PCI Study. JACC Cardiovasc Interv. 2019 Oct 28;12(20):1991-2001. doi: 10.1016/j.jcin.2019.05.054. PMID 31648761
- [Background] Tebaldi M, Biscaglia S, Fineschi M, Musumeci G, Marchese A, Leone AM, Rossi ML, Stefanini G, Maione A, Menozzi A, Tarantino F, Lodolini V, Gallo F, Barbato E, Tarantini G, Campo G. Evolving Routine Standards in Invasive Hemodynamic Assessment of Coronary Stenosis: The Nationwide Italian SICI-GISE Cross-Sectional ERIS Study. JACC Cardiovasc Interv. 2018 Aug 13;11(15):1482-1491. doi: 10.1016/j.jcin.2018.04.037. Epub 2018 May 23. PMID 29803695
- [Background] Piroth Z, Toth GG, Tonino PAL, Barbato E, Aghlmandi S, Curzen N, Rioufol G, Pijls NHJ, Fearon WF, Juni P, De Bruyne B. Prognostic Value of Fractional Flow Reserve Measured Immediately After Drug-Eluting Stent Implantation. Circ Cardiovasc Interv. 2017 Aug;10(8):e005233. doi: 10.1161/CIRCINTERVENTIONS.116.005233. PMID 28790165
- [Derived] Marrone A, Erriquez A, Verardi FM, Colaiori I, Cocco M, Caglioni S, Tumscitz C, Penzo C, Marchini F, Meinen J, McNutt J, Buijs JOD, Chiu WC, Versaci F, Campo G, Biscaglia S. Additional Value of Optical Coherence Tomography-Derived Virtual Flow Reserve for Percutaneous Coronary Intervention Guidance. Catheter Cardiovasc Interv. 2025 Dec;106(7):3456-3464. doi: 10.1002/ccd.70207. Epub 2025 Sep 23. PMID 40988408
- [Derived] Biscaglia S, Verardi FM, Tebaldi M, Guiducci V, Caglioni S, Campana R, Scala A, Marrone A, Pompei G, Marchini F, Scancarello D, Pignatelli G, D'Amore SM, Colaiori I, Demola P, Di Serafino L, Tumscitz C, Penzo C, Erriquez A, Manfrini M, Campo G. QFR-Based Virtual PCI or Conventional Angiography to Guide PCI: The AQVA Trial. JACC Cardiovasc Interv. 2023 Apr 10;16(7):783-794. doi: 10.1016/j.jcin.2022.10.054. Epub 2023 Mar 8. PMID 36898939